CLINICAL TRIAL: NCT05827263
Title: Temporary Hydrostatic Splint Therapy and Its Effects on Occlusal Forces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Gediminas Žekonis, Professor, Lithuanian University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BE-2-48
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Occlusal splints; Dental occlusion; Balanced Dental Occlusion; Temporomandibular Joint Disorders; Bite Force; Centric Dental Occlusion; Dental Equipment
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bites and Stings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group - non-temporomandibular disorders group. (Active Comparator): Patients diagnosed with no temporomandibular disorders.
  Interventions: Diagnostic Test: T-Scan occlusal recording No. I; Device: Usage of the hydrostatic appliance; Diagnostic Test: T-Scan occlusal recording No. II
- Test group - temporomandibular disorders group (Experimental): Patients diagnosed with mild, moderate, or severe temporomandibular disorders.
  Interventions: Diagnostic Test: T-Scan occlusal recording No. I; Device: Usage of the hydrostatic appliance; Diagnostic Test: T-Scan occlusal recording No. II

INTERVENTIONS:
Diagnostic Test: T-Scan occlusal recording No. I — Occlusal information was obtained using the T-Scan device before the main intervention. This process was repeated three times to confirm the findings.
Device: Usage of the hydrostatic appliance — The hydrostatic appliance was removed from its packaging and placed symmetrically between the upper lip and the oral vestibule of the maxilla for the most comfortable position. After 30 minutes, the hydrostatic appliance was removed, and patients were asked to keep their mouths open until the T-Scan was positioned correctly.
Diagnostic Test: T-Scan occlusal recording No. II — The occlusal registration was repeated three times using the T-Scan device in order to confirm the findings.

SUMMARY:
The goal of this non-randomized controlled trial is to analyze and compare occlusal force distribution patterns using T-Scan III before and after hydrostatic splint therapy on both healthy subjects and subjects with temporomandibular disorders. The main questions it aims to answer are:

* Do occlusal forces for individual teeth differ before and after hydrostatic splint therapy?
* Does the percentage distribution of forces across different sectors differ before and after hydrostatic splint therapy?

Participants will:

* Perform occlusal analysis using the T-Scan III device;
* Use a hydrostatic splint for 30 minutes;
* Perform a second occlusal analysis after using the hydrostatic splint.

Researchers will compare healthy subjects and subjects with temporomandibular disorders to see if hydrostatic splint therapy makes a difference in the distribution patterns of occlusal forces.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects with Angle Class I and a normal line of occlusion without malpositioned or rotated teeth;
* complete permanent dentition except for the third molars;
* no fixed prosthesis;
* no dental caries;
* no restorations on the occlusal surfaces of molars and premolars extending more than one-third of the surface;
* no restorations on incisal edge;
* no tenderness on percussion of any teeth;
* no history of previous endodontic and orthodontic treatment,
* extensive maxillofacial surgery;
* no systematic neurological disorders.

Exclusion Criteria:

* presence of orofacial pain that limits mouth opening;
* malocclusion (e.g., open bite, increased overjet or reverse overjet, cross bite);
* skeletal anomalies with occlusal disturbance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change of percentage force distribution per sector. | Change of percentage force distribution per sector at 30-minute of hydrostatic appliance usage.
Change of percentage force distribution for single dental elements. | Change of percentage force distribution for single dental elements at 30-minute of hydrostatic appliance usage.

CONTACTS AND LOCATIONS:
Overall Officials: Mante Kireilyte, Study Chair — Lithuanian University of Health Sciences
Locations (1):
- MK Dental Studio, Marijampolė, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Yes, there is a plan to make individual participant data and related data dictionaries available to other researchers. In addition to sharing the individual participant data, we also plan to publish a scientific article in the Journal of Dental Research to disseminate our findings.